CLINICAL TRIAL: NCT05759442
Title: Clinical Efficacy and Safety of Metformin Versus Apple Cider Vinegar (ACV) in Prediabetics
Acronym: BUHSCK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Dr. Shizma Junejo, Senior Lecturer Pharmacology Department, Bahria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERC 123/2022
Record Dates: First submitted 2023-02-18; First posted 2023-03-08 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: PreDiabetes
Keywords: Prediabetes; Metformin HCl; Apple cider vinegar
MeSH Terms: conditions — Prediabetic State | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Randomized, open label, prospective, clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Active Comparator): Tablet Metformin HCl 500 mg per oral twice daily for 12 weeks
  Interventions: Drug: Metformin Hydrochloride (HCL)
- Apple cider vinegar (Active Comparator): Apple Cider Vinegar 15ml per day diluted in 200 ml of water for 12 weeks
  Interventions: Dietary Supplement: Apple cider vinegar

INTERVENTIONS:
Drug: Metformin Hydrochloride (HCL) — Tab Metformin HCL 500mg twice per day aimed at improving glycemic indices in Prediabetics
  Arms: Metformin
Dietary Supplement: Apple cider vinegar — Apple cider vinegar aimed at improving glycemic indices in Prediabetics
  Arms: Apple cider vinegar

SUMMARY:
The goal of this clinical trial is to compare efficacy and safety of metformin versus apple cider vinegar in prediabetics . The main question[s] it aims to answer are:

* Efficacy of metformin versus apple cider vinegar in prediabetics
* Safety of metformin versus apple cider vinegar in prediabetics

Researchers will compare group of prediabetics taking metformin with group of prediabetics taking apple cider vinegar to see if there is difference in safety and efficacy..

ELIGIBILITY:
Inclusion Criteria:

* Males and Female
* 17-40 years age
* Body Mass index (BMI) overweight and obese
* FBS (100-125 mg/dl)
* HBA1c 5.7% to 6.4%

Exclusion Criteria:

* Concomitant medical problems as established diabetes, hepatic or renal insufficiencies etc.
* Known allergy or intolerance to metformin or apple cider vinegar

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Glycated Hemoglobin | 12 weeks
  Change in glycosylated hemoglobin (HbA1c ) in percent
Fasting Blood Sugar | 12 weeks
  Change in fasting blood sugar (FBS) in mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Shizma Junejo, MBBS,MSc, Principal Investigator — Bahria University Health Sciences Campus
Locations (1):
- Diabetologist Clinics (02), Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No